CLINICAL TRIAL: NCT05443074
Title: Efficacy of a Face-to-face Versus a Remote Physiotherapy Instruction Session About Pelvic Floor in the Pelvic Floor Muscle Capacity of Incontinent Women: a Randomized Controlled Trial
Brief Title: Efficacy of a Face to Face Versus a Remote Physiotherapy Instruction Session About Pelvic Floor in Women With Urinary Incontinence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Caroline Caetano Pena, Principal investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 52672521.0.0000.5440
Record Dates: First submitted 2022-05-24; First posted 2022-07-05 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Face to face intervention group (Active Comparator): This group will be composed of participants who will receive face to face physiotherapy instruction session.
  Interventions: Other: Face to face intervention group
- Remote intervention group (Experimental): This group will be composed of participants who will receive real time remote physiotherapy instruction session.
  Interventions: Other: Remote intervention group
- Control group (Active Comparator): This group will be composed of participants who will not receive any type of physiotherapy instruction session during the period of the study.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Face to face intervention group — Participants of this group will participate in a one 15 minutes face to face session where they will receive information about anatomy, functions and dysfunctions of the pelvic floor. During the session, some teaching materials will be used (an anatomical model, prototype simulator of the functions of the PFM, posters, videos and images), in order to facilitate the learning of women about how to contract their PFM and how to avoid urinary loss by contracting their muscles.
  At the end of the session, the participants will have time to ask their questions and will receive a home booklet reinforcing the information given during the session including instructions for them to perform a PFM contraction during daily live situations that generate an increased intra-abdominal pressure, such as coughing, sneezing, weight lifting and other activities, as well as strategies to inhibit urge urinary incontinence (UI).
  Arms: Face to face intervention group
Other: Remote intervention group — Participants of this group will be referred to a room with a computer (inside the rehabilitation center) to participate in a one 15 minutes real time remote session, where they will receive information about anatomy, functions and dysfunctions of the pelvic floor. During the session, some teaching materials will be used (an anatomical model, prototype simulator of the functions of the PFM, posters, videos and images), in order to facilitate the learning of women about how to contract their PFM and how to avoid urinary loss by contracting their muscles.
  At the end of the session, the participants will have time to ask their questions and will receive a home booklet reinforcing the information given during the session including instructions for them to perform a PFM contraction during daily live situations that generate an increased intra-abdominal pressure, such as coughing, sneezing, weight lifting and other activities, as well as strategies to inhibit urge UI.
  Arms: Remote intervention group
Other: Control group — Participants of this group will be assessed in the same time points of the participants of the two other groups. They will not receive any intervention or information about pelvic floor anatomy, functions and dysfunctions of the pelvic floor, however after the last assessment (20 days after) for ethical reasons they will receive the same intervention.
  Arms: Control group

SUMMARY:
The purpose of this study is to assess and to compare the efficacy of a face to face versus a remote physiotherapy instruction session about pelvic floor muscle (PFM) function, including teaching women how to contract their PFM and how to perceive a correct PFM contraction. Study participants will be randomly assigned to participate in one of the three study groups: Group 1 will receive face to face instructions, Group 2 will receive real time remote instructions and Group 3 will not receive any instruction. The primary outcome measure is PFM function assessed using the modified Oxford Scale.

ELIGIBILITY:
Inclusion Criteria:

* Women who are not able to contract their PFM (≤ 2 of Modified Oxford Scale);
* Cognitive ability, hearing and visual acuity preserved (through 10-point cognitive screener and Snellen test, respectively);
* Non-neurogenic UI;
* No history of neurological disorders;
* No symptoms of a vaginal or urinary tract infection;
* Pelvic organ prolapse ≤2 (according to the Baden and Walker scale);
* Who have not already been instructed on how to perform PFM contraction or who is not already performing PFM training;
* No suspected or confirmed pregnancy.

Exclusion Criteria:

* Who have intolerance to physical examination, or latex allergy;
* Who withdraws from participating in the study.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Change in contraction capacity | At baseline, immediately after intervention and 20 days after the intervention.
  The Modified Oxford Scale will be used to assess change in the capacity to perform a PFM contraction through vaginal palpation. The Modified Oxford Scale is a categorical variable with 6 possible answers ranging from 0 to 5. High scores of Modified Oxford Scale mean better PFM function and lower scores mean worse PFM function.
Change in self-perception of the PFM | At baseline, immediately after intervention and 20 days after the intervention.
  The Modified Oxford Scale will be used to assess change in the participants' self-perception of their contraction after vaginal palpation. The Modified Oxford Scale is a categorical variable with 6 possible answers ranging from 0 to 5. High scores of Modified Oxford Scale mean better PFM function and lower scores mean worse PFM function.

SECONDARY OUTCOMES:
Self-report of UI symptoms | At baseline and 20 days after the intervention.
  Reports of UI symptoms will be evaluated through the International Consultation on Incontinence Questionnaire - Short Form. Participants who report having had no urinary leakage in the last four weeks will be considered continents. The International Consultation on Incontinence Questionnaire score can range from 0 (when there is no report of urinary leakage, with no impact on quality of life) to 21 (highest in UI severity and maximum impact on quality of life).
Assessment of the usefulness of teaching resources | Immediately after intervention
  The usefulness of teaching resources will be evaluated by the numerical visual scale and by a questionnaire developed by the researchers. In the post-intervention evaluation of face to face intervention group and remote intervention group, the numerical visual scale and the questionnaire will be presented to the participants and then they will be asked to evaluate and mark on the line the point corresponding to the degree of satisfaction/usefulness of the resources. Scores closer to 0 correspond to no satisfaction with the resources used in the instruction session about pelvic floor and scores closer to 10 correspond to satisfaction with the resources used.
Satisfaction with the orientations | Immediately after intervention
  Satisfaction with the instructions received during the session will be evaluated by the numerical visual scale. In the post-intervention evaluation, face to face intervention group and remote intervention group will be asked to evaluate and mark on the line the point corresponding to the degree of satisfaction with the guidelines given in the session. Scores closer to 0 correspond to no satisfaction with the instruction received during session about pelvic floor and scores closer to 10 correspond to satisfaction with the instruction received during session about pelvic floor.
System usability assessment | Immediately after intervention
  The usability of the system used to carry out the remote intervention group session will be evaluated through the systems usability scale. The system usability assessment score can range from 0 (the lower the score, the greater the usability problems of the system used) to 100 (the higher the score, the lower the usability problems of the system used).

CONTACTS AND LOCATIONS:
Overall Officials: Cristine H Jorge, Study Director — University of Sao Paulo
Locations (1):
- University of São Paulo, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aoki Y, Brown HW, Brubaker L, Cornu JN, Daly JO, Cartwright R. Urinary incontinence in women. Nat Rev Dis Primers. 2017 Jul 6;3:17042. doi: 10.1038/nrdp.2017.42. PMID 28681849
- [Background] Bo K, Frawley HC, Haylen BT, Abramov Y, Almeida FG, Berghmans B, Bortolini M, Dumoulin C, Gomes M, McClurg D, Meijlink J, Shelly E, Trabuco E, Walker C, Wells A. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for the conservative and nonpharmacological management of female pelvic floor dysfunction. Neurourol Urodyn. 2017 Feb;36(2):221-244. doi: 10.1002/nau.23107. Epub 2016 Dec 5. PMID 27918122
- [Background] Cacciari LP, Dumoulin C, Hay-Smith EJ. Pelvic floor muscle training versus no treatment, or inactive control treatments, for urinary incontinence in women: a cochrane systematic review abridged republication. Braz J Phys Ther. 2019 Mar-Apr;23(2):93-107. doi: 10.1016/j.bjpt.2019.01.002. Epub 2019 Jan 22. PMID 30704907
- [Background] Dantas LO, Barreto RPG, Ferreira CHJ. Digital physical therapy in the COVID-19 pandemic. Braz J Phys Ther. 2020 Sep-Oct;24(5):381-383. doi: 10.1016/j.bjpt.2020.04.006. Epub 2020 May 1. No abstract available. PMID 32387004
- [Background] de Andrade RL, Bo K, Antonio FI, Driusso P, Mateus-Vasconcelos ECL, Ramos S, Julio MP, Ferreira CHJ. An education program about pelvic floor muscles improved women's knowledge but not pelvic floor muscle function, urinary incontinence or sexual function: a randomised trial. J Physiother. 2018 Apr;64(2):91-96. doi: 10.1016/j.jphys.2018.02.010. Epub 2018 Mar 21. PMID 29574170
- [Background] de Freitas LM, Bo K, Fernandes ACNL, Uechi N, Duarte TB, Ferreira CHJ. Pelvic floor muscle knowledge and relationship with muscle strength in Brazilian women: a cross-sectional study. Int Urogynecol J. 2019 Nov;30(11):1903-1909. doi: 10.1007/s00192-018-3824-y. Epub 2018 Nov 22. PMID 30467764
- [Background] Ferreira CHJ, Driusso P, Haddad JM, Pereira SB, Fernandes ACNL, Porto D, Reis BM, Mascarenhas LR, Brito LGO, Ferreira EAG. A guide to physiotherapy in urogynecology for patient care during the COVID-19 pandemic. Int Urogynecol J. 2021 Jan;32(1):203-210. doi: 10.1007/s00192-020-04542-8. Epub 2020 Sep 28. PMID 32986147
- [Background] Fernandes ACNL, Palacios-Cena D, Hay-Smith J, Pena CC, Sidou MF, de Alencar AL, Ferreira CHJ. Women report sustained benefits from attending group-based education about pelvic floor muscles: a longitudinal qualitative study. J Physiother. 2021 Jul;67(3):210-216. doi: 10.1016/j.jphys.2021.06.010. Epub 2021 Jun 17. PMID 34147398
- [Background] Frawley HC, Galea MP, Phillips BA, Sherburn M, Bo K. Reliability of pelvic floor muscle strength assessment using different test positions and tools. Neurourol Urodyn. 2006;25(3):236-242. doi: 10.1002/nau.20201. PMID 16299815
- [Background] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Int Urogynecol J. 2010 Jan;21(1):5-26. doi: 10.1007/s00192-009-0976-9. Epub 2009 Nov 25. PMID 19937315
- [Background] Hay-Smith J, Herderschee R, Dumoulin C, Herbison P. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women: an abridged Cochrane systematic review. Eur J Phys Rehabil Med. 2012 Dec;48(4):689-705. PMID 23183454
- [Background] Hui E, Lee PS, Woo J. Management of urinary incontinence in older women using videoconferencing versus conventional management: a randomized controlled trial. J Telemed Telecare. 2006;12(7):343-7. doi: 10.1258/135763306778682413. PMID 17059650
- [Background] Laycock J. Pelvic muscle exercises: physiotherapy for the pelvic floor. Urol Nurs. 1994 Sep;14(3):136-40. No abstract available. PMID 7732416
- [Background] Liao YM, Dougherty MC, Liou YS, Tseng IJ. Pelvic floor muscle training effect on urinary incontinence knowledge, attitudes, and severity: an experimental study. Int J Nurs Stud. 2006 Jan;43(1):29-37. doi: 10.1016/j.ijnurstu.2005.01.004. PMID 16326162
- [Background] Mateus-Vasconcelos ECL, Brito LGO, Driusso P, Silva TD, Antonio FI, Ferreira CHJ. Effects of three interventions in facilitating voluntary pelvic floor muscle contraction in women: a randomized controlled trial. Braz J Phys Ther. 2018 Sep-Oct;22(5):391-399. doi: 10.1016/j.bjpt.2017.12.006. Epub 2018 Feb 3. PMID 29429823
- [Background] Miller JM, Ashton-Miller JA, DeLancey JO. A pelvic muscle precontraction can reduce cough-related urine loss in selected women with mild SUI. J Am Geriatr Soc. 1998 Jul;46(7):870-4. doi: 10.1111/j.1532-5415.1998.tb02721.x. PMID 9670874
- [Background] Nelson ME, Rejeski WJ, Blair SN, Duncan PW, Judge JO, King AC, Macera CA, Castaneda-Sceppa C. Physical activity and public health in older adults: recommendation from the American College of Sports Medicine and the American Heart Association. Med Sci Sports Exerc. 2007 Aug;39(8):1435-45. doi: 10.1249/mss.0b013e3180616aa2. PMID 17762378
- [Background] Scott Kruse C, Karem P, Shifflett K, Vegi L, Ravi K, Brooks M. Evaluating barriers to adopting telemedicine worldwide: A systematic review. J Telemed Telecare. 2018 Jan;24(1):4-12. doi: 10.1177/1357633X16674087. Epub 2016 Oct 16. PMID 29320966
- [Background] Smith AL, Nissim HA, Le TX, Khan A, Maliski SL, Litwin MS, Sarkisian CA, Raz S, Rodriguez LV, Anger JT. Misconceptions and miscommunication among aging women with overactive bladder symptoms. Urology. 2011 Jan;77(1):55-9. doi: 10.1016/j.urology.2010.07.460. Epub 2010 Oct 23. PMID 20970839
- [Background] Talasz H, Himmer-Perschak G, Marth E, Fischer-Colbrie J, Hoefner E, Lechleitner M. Evaluation of pelvic floor muscle function in a random group of adult women in Austria. Int Urogynecol J Pelvic Floor Dysfunct. 2008 Jan;19(1):131-5. doi: 10.1007/s00192-007-0404-y. Epub 2007 Sep 18. PMID 17876492
- [Background] Tibaek S, Dehlendorff C. Pelvic floor muscle function in women with pelvic floor dysfunction: a retrospective chart review, 1992-2008. Int Urogynecol J. 2014 May;25(5):663-9. doi: 10.1007/s00192-013-2277-6. Epub 2013 Dec 12. PMID 24337586
- [Background] Uechi N, Fernandes ACNL, Bo K, de Freitas LM, de la Ossa AMP, Bueno SM, Ferreira CHJ. Do women have an accurate perception of their pelvic floor muscle contraction? A cross-sectional study. Neurourol Urodyn. 2020 Jan;39(1):361-366. doi: 10.1002/nau.24214. Epub 2019 Nov 18. PMID 31737927
- [Derived] Hay-Smith EJC, Starzec-Proserpio M, Moller B, Aldabe D, Cacciari L, Pitangui ACR, Vesentini G, Woodley SJ, Dumoulin C, Frawley HC, Jorge CH, Morin M, Wallace SA, Weatherall M. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2024 Dec 20;12(12):CD009508. doi: 10.1002/14651858.CD009508.pub2. PMID 39704322